CLINICAL TRIAL: NCT04967690
Title: An Open-label Dose Escalation Study to Estimate MTD, Identify DLTs and Study Pharmacokinetics Following a Single Dose of Intracranially Administered Temozolomide-based SI-053 as an add-on to the Current Standard of Care, in Adult Patients With Newly Diagnosed Glioblastoma
Brief Title: A Dose Escalation Study to Estimate MTD, DLTs and Pharmacokinetics After a Single Intracranial Dose of SI-053 as an add-on to the Current Standard of Care, in Adult Patients With Newly Diagnosed GBM
Acronym: TARGLIO
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Double Bond Pharmaceutical AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DBP-053-01
Record Dates: First submitted 2021-06-30; First posted 2021-07-19 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Newly Diagnosed Glioblastoma

STUDY DESIGN:
Intervention Model Description: Up to 27 subjects will be included in the trial (estimated; 21 subjects in total for dose escalation following a 3+3 rule based design for six doses in total, including three more subjects at RP2D, and an additional six subjects for dose expansion at RP2D).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SI-053 (Experimental): Single arm study. Dose escalation will follow a rule-based 3 + 3 design using increasing doses of SI-053. Subjects will receive a single i.c. dose of room-tempered SI-053 gel, which will be applied onto the walls of the cavity formed after tumor resection using a sterile spatula.This will be followed by chemo-radiotherapy commencing at least 21 and no later than 35 days after SI-053 administration. The dose escalation part of the trial will follow a rule-based 3 + 3 design using a total of six dose levels of SI-053 (optional dose of 50 mg will be used to de-escalate in case of DLT at 75 mg) that consist of increasing amounts of TMZ in a constant amount of excipient and sterile WFI. These dose levels are planned to be tested in 21 subjects, including three more subjects at preliminary RP2D.The dose expansion phase will enroll an additional six subjects,to be treated at the RP2D in order to gather additional safety and preliminary efficacy data at that dose.
  Interventions: Drug: SI-053

INTERVENTIONS:
Drug: SI-053 — SI-053 will be used as an add-on to SoC for newly diagnosed GBM.In conjunction with surgical resection, SI-053 will be applied intracranially (i.c.) into the cavity that is formed after tumor resection. Post-operative chemoradiotherapy (including concomitant and adjuvant TMZ or following the CeTeG protocol) will be initiated at least 21 and no later than 35 days after SI-053 administration.

SUMMARY:
SI-053 is a novel powder formulation containing temozolomide (TMZ), an alkylating chemotherapy agent, in an excipient which forms a viscous gel upon reconstitution in water. SI-053 will be used as an add-on to SoC for newly diagnosed GBM. SoC consists of maximal safe resection followed by radiation therapy (RT) with concomitant TMZ and adjuvant chemotherapy with TMZ. For MGMT promoter methylated GBM, lomustine and TMZ may be administered plus radiation therapy

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF) prior to the start of any trial-related procedures.
2. Subject age ≥ 18 years with an upper limit of 70 years.
3. In the Investigator's opinion, subject is able and willing to comply with all trial requirements for the duration of the trial.
4. Suspected primary, newly diagnosed supratentorial GBM (Grade IV glioma per WHO guidelines) based on signs/symptoms and MRI (obtained maximally 10 days prior to surgery, using the same MRI settings as will be used for post-surgery MRI; if the MRI is older than 10 days or if it is taken at a local clinic, this has to be repeated within 10 days before the surgery), needing maximum safe resection followed by chemoradiotherapy as per institutional guidelines (Stupp protocol: radiotherapy [60 Gy total; 10 Gy per week for 6 weeks] plus concomitant TMZ [75 mg/m2 of body surface area per day; 7 days per week from first to the last day of radiotherapy], followed by six cycles of adjuvant TMZ [150 to 200 mg/m2] once daily for 5 consecutive days, followed by 23 days of no treatment prior to the next cycle; or CeTeG protocol for MGMT promoter methylated GBMs: up to six courses of lomustine [100 mg/m2 on Day 1 plus TMZ [100-200 mg/m2 per day on Days 2-6 of the 6-week course] in addition to radiotherapy [59-60 Gy], if preferred by the investigator).
5. Preliminary histological diagnosis of GBM by an intraoperative "frozen section", analyzed during surgery is mandatory before administration of SI-053. A final diagnosis is made by histopathological and molecular analysis of the resected tumor tissue.
6. It is the surgeon's estimation that maximum safe resection of the contrast enhancing part of the tumor with image-guided surgery is possible and it is not expected that the ventricular system will be opened during surgery. When the ventricular system is opened during surgery, no SI-053 will be administered.
7. The tumor volume as assessed by pre-surgery MRI is at least 10 mL, and the actual resection bed volume based on the surgeon's estimation after surgery enables complete administration of a single dose of SI-053.
8. Karnofsky Performance Status (KPS) score ≥70%
9. Women of childbearing potential (WOCBP) and men whose partner is of childbearing potential must use effective contraception from the time of screening and for 6 months after receiving SI-053. WOCBP should have a negative serum pregnancy test β-human chorionic gonadotropin (β-HCG) at trial enrollment and within ≤ 72 h before SI-053 administration.
10. Subjects must have following laboratory values obtained within 2 weeks prior to enrollment.

    • Acceptable liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (except in the case of Gilbert's disease); Albumin 3.0 - 5.5 g/dL; Aspartate transaminase (AST) ≤ 2.5 x ULN
    * Alanine transaminase (ALT) ≤ 2.5 x ULN
    * Alkaline phosphatase ≤ 2.5 x ULN
    * Acceptable kidney function: Creatinine clearance: ≤ 30 mL/min (by CKD-EPI formula)
    * Acceptable hematologic status:

    Absolute neutrophil count (ANC) ≥ 1 500 cells/mm3 Platelet count ≥ 100 000 cells/mm3 Hemoglobin ≥ 10.0 g/dL
11. Subjects should have a suspected life expectancy of at least 6 months.
12. Documented negative test for HBV. For HBV serology, the determination of hBsAg and anti-hBcAg Ab is required.

Exclusion Criteria:

* Subjects who fulfil any of the following criteria will be excluded from the trial:

  1. Prior treatment for GBM including resection or radiation therapy.
  2. Contraindications to radiation therapy or TMZ chemotherapy (i.e allergy, hypersensitivity or other intolerabilities to TMZ and its excipients or hypersensitivity to dacarbazine).
  3. Has a history of another primary malignancy, except for:

     * Malignancy treated with curative intent and with no known active disease within 2 years prior to SI-053 administration
     * Adequately treated non-invasive basal skin cancer or squamous cell skin carcinoma
     * Adequately treated uterine cervical cancer stage 1B or less
  4. Has clinically significant cardiac disease (as identified by electrocardiogram [ECG]), including:

     * Known congestive heart failure Grade III or IV by the New York Heart Failure Association;
     * Myocardial infarction within 6 months prior to signing the ICF;
     * Onset of unstable angina within 6 months prior to signing the ICF.
  5. Infratentorial or multifocal glioblastoma.
  6. Pre-operative MRI showing ventricular invasion (defined as presence of intraventricular lesion or of intraventricular tumor mass).
  7. Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1.
  8. Chronic use of systemic steroid therapy (>1 month of >10 mg prednisone per day or equivalent, except topical or inhaled).
  9. Any significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or affect the participant's ability to participate in the trial.
  10. Subjects who have participated in another research trial involving an investigational product within the past 12 weeks or are currently participating in another clinical trial (excluding observational studies).
  11. Pregnant or lactating women.
  12. Subjects unable to undergo MRI during the trial participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence rate and the grade (severity) of dose-limiting toxicities (DLTs) of a single i.c dose of SI-053 | 6 months
  • Incidence rate and the grade (severity) of dose-limiting toxicities (DLTs) based on the occurrence of adverse events (AEs) reported according to the National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE) v 5.0
SI-053 related adverse events (AEs) and toxicity | 6 months
  SI-053 related AEs and toxicity determined by evaluation of the extent of edema (and associated use of steroids to control edema), neurological toxicities (e.g. sudden increase in seizure activity as a result of local inflammation), any infection (by requirement for antibiotic treatment), additional surgery or any additional treatment that would delay the chemoradiotherapy.

SECONDARY OUTCOMES:
Determination of plasma concentration of TMZ and its metabolite 5-amino-1H-imidazole-4-carboxamide (AIC) and PK parameters | 6 months
  Determination of plasma concentration of TMZ and its metabolite 5-amino-1H-imidazole-4-carboxamide (AIC) and PK parameters

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Westphal, Prof.Dr.Med., Principal Investigator — Universitätklinikum Hamburg-Eppendorf, Martinistrasse 52, 20246 Hamburg, Germany